CLINICAL TRIAL: NCT01577615
Title: Patterned Experience for Preterm Infants
Acronym: PEPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NR012307-02 (NIH)
Record Dates: First submitted 2012-04-11; First posted 2012-04-16 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Complication of Prematurity
Keywords: Preterm Infant; Neurobehavioral; Development
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patterned Experience Group (Experimental): Infants in the patterned experience group will receive a patterned feeding experience with all feedings through discharge. They will receive a touch intervention at each gavage feeding. Once oral feedings are initiated, they will be offered an oral feeding at every scheduled feeding. They will be held for feedings. They will be observed twice a week utilizing the computer data acquisition system. Follow up visits will occur at 2,6 amd 24 months corrected age.
  Interventions: Behavioral: Patterned Experience
- Usual Care Group (No Intervention): In the usual care group infants usually are not held or contained during gavage feeding. Infants in the usual care group are orally fed at the discretion of the nurses or medical team. Once oral feedings are initiated, infants will be observed twice a week using the computer data acquisition system. Follow up visits will occur at 2,6 and 24 months corrected age.

INTERVENTIONS:
Behavioral: Patterned Experience — * The caregiver's hand over the shoulder area and the other hand over the lower extremities during feeding in the incubator, swaddling or holding outside the incubator.
  * Nonnutritive sucking will be offered to infants.
  * Blood work will be collected for inflammatory cytokines.
  * Saliva will be collected for genetic analysis
  * Saliva will be collected in 10 infant sub study for cortisol pre and post feedings
  * All scheduled feedings will include an opportunity for the infant to try feeding orally by bottle or breast while being held in a swaddled flexed position.
  * Once bottle feedings are initiated, infants will be observed twice a week utilizing the computer data acquisition system.
  * Follow up visits will occur at 2,6and 24 months corrected age.
  Arms: Patterned Experience Group

SUMMARY:
The PEPI study is designed to provide a patterned feeding experience. By using a regularly occurring and necessary caregiving event, feeding, as the vehicle for the patterned experience, the intervention should be effective at promoting and reinforcing neuronal growth and connections that are critical for neurobehavioral and cognitive function while at the same time being cost effective in its delivery.

DETAILED DESCRIPTION:
Infants will be randomly assigned to a study group or control group. The research study will last for approximately twenty four months. Infants will have daily assessments while in the hospital and three study visits after hospital discharge. All post-discharge visits will occur in an out patient hospital setting. During the first days of life, study staff will start observing infant's development by using assessment tools. Lab samples include one blood sample taken when other blood is being collected in the first days of life and one saliva sample when the infants starts bottle feeding.

When tube feedings are started in the study group, caregivers (nurses, parents or research staff) will gently place hands on the infant while in the incubator (ill babies) or bundled outside the incubator. If the infant is in the control group, they will receive standard tube feeding care.

When oral feedings are started in the study group, the infant will have an opportunity at every feeding to be breast or bottle fed while being held. If unable to complete the entire feeding orally, the rest will be tube fed.

If the infant is in the control group, feeding opportunities will be decided by the medical team providing care.

All infants will be observed during oral feedings twice a week while in the hospital. Study staff will watch heart rate, sucking activity (a sensor on the chin) and level of wakefulness.

ELIGIBILITY:
Inclusion Criteria:

* Infants born ≤ 32 weeks gestation

Exclusion Criteria:

* Infants will be excluded if the infant has gastrointestinal, craniofacial, cardiovascular, neuromuscular, and/or genetic defects

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Neurobehavioral Assessment of the Preterm Infant (NAPI) | Birth, Transition to by mouth feeding, hospital discharge, 2 mo corrected age
  Used as a measure of neurobehavioral development.

SECONDARY OUTCOMES:
Bailey Scale of Infant Development (BSID), 3rd edition | 6 and 24 months corrected age
  Used as a measure of cognitive development.
Sucking activity | Changes from an average age of 33 weeks postmenstural age to an average age of 38 weeks postmenstural age.
  Used as a measure of central nervous system organization once oral feeding is initiated.
Heart rate variability (low frequency:high frequency ratio) | Changes from an average age of 33 weeks postmenstural age to an average age fo 38 weeks postmenstural age.
  Used as a measure of autonomic system organization once oral feedings are initiated.

CONTACTS AND LOCATIONS:
Overall Officials: Rita H Pickler, PhD, RN, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - University of Cincinnati Health Center, Cincinnati, Ohio
  - Cincinnati Children's Medical Center, Cincinnati, Ohio

REFERENCES:
- [Derived] Pickler RH, Meinzen-Derr J, Moore M, Sealschott S, Tepe K. Effect of Tactile Experience During Preterm Infant Feeding on Clinical Outcomes. Nurs Res. 2020 Sep/Oct;69(5S Suppl 1):S21-S28. doi: 10.1097/NNR.0000000000000453. PMID 32555011
- [Derived] Nist MD, Shoben AB, Pickler RH. Early Inflammatory Measures and Neurodevelopmental Outcomes in Preterm Infants. Nurs Res. 2020 Sep/Oct;69(5S Suppl 1):S11-S20. doi: 10.1097/NNR.0000000000000448. PMID 32496397
- [Derived] Pickler R, Sealschott S, Moore M, Merhar S, Tkach J, Salzwedel AP, Lin W, Gao W. Using Functional Connectivity Magnetic Resonance Imaging to Measure Brain Connectivity in Preterm Infants. Nurs Res. 2017 Nov/Dec;66(6):490-495. doi: 10.1097/NNR.0000000000000241. PMID 29095379
- [Derived] Pickler RH, Wetzel PA, Meinzen-Derr J, Tubbs-Cooley HL, Moore M. Patterned feeding experience for preterm infants: study protocol for a randomized controlled trial. Trials. 2015 Jun 4;16:255. doi: 10.1186/s13063-015-0781-3. PMID 26041365